CLINICAL TRIAL: NCT04888598
Title: Study of the Microvascular Changes in the Retina Measured by Optical Coherence Tomography (OCT) - Angiography in Patients With Type 1 Diabetes Mellitus at the Onset of the Disease and After Optimization of Glycemic Control.
Brief Title: Microvascular Changes in OCT-angiography in Type 1 Diabetes Mellitus at the Onset of the Disease and After Optimization of Glycemic Control.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Arnau de Vilanova (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-RET-2020-69
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Type 1 Diabetes; Diabetic Retinopathy
Keywords: OCT-A; OCT Angiography
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Retinopathy | interventions — Tomography, Optical Coherence; Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Type 1 diabetic patients: Recently diagnosed type 1 diabetes patients
  Interventions: Diagnostic Test: Optical Coherence Tomography (OCT) Angiography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography (OCT) Angiography — Measurement of retinal vessel density and distribution in the macula using new generation OCT device

SUMMARY:
The objective of the study is to evaluate the differences in the retinal microcirculation measured by OCT-Angiography in patients with type 1 diabetes between the diagnosis of the disease and after 3 months of insulin treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 Diabetes at diagnosis of the disease (less than 7 days after diagnosis)
* Age equal to or greater than 18 years
* Signature of the informed consent by the patient / legal guardian.

Exclusion Criteria:

* Metabolic situation of ketosis or ketoacidosis, according to clinical criteria established in the protocol of the Endocrinology and Nutrition Service. The patient will be a candidate once the ketonemia is absent (value <1 mmol / L).
* Previous diagnosis of dyslipidemia and any previous lipid-lowering treatment
* Previous diagnosis of hypertension and any previous hypotensive treatment
* Previous diagnosis of any form of cardiovascular disease, including heart failure.
* Previous kidney disease, and presence of advanced kidney failure (estimated glomerular filtration rate <60 ml / min)
* Presence of diabetic retinopathy identifiable by conventional eye fundus or retinography, or other concomitant retinal vascular pathology (hypertensive retinopathy, venous occlusion, arterial obstruction, etc.)
* History or presence of retinal pathology that may alter its structure and / or the validity of the measurements (retinal detachment, epiretinal membrane, high myopia -understood as an axial length greater than or equal to 26mm measured by "IOL Master" biometry-, neovascular membrane, choroidal tumors, etc.)
* History of posterior uveitis or retinal vasculitis
* Glaucoma and neuro-ophthalmological pathology that can alter the neuroretinal structures.
* Refractive media opacity that prevents a correct acquisition of images and, therefore, their evaluation
* Dementia or intellectual disability that prevent proper collaboration when acquiring images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with type 1 diabetes who meet all the inclusion criteria and none of the exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Vessel density | 3 months
  Density of retinal vessels and perfusion in the macula

SECONDARY OUTCOMES:
Vessel density | 6 months
  Density of retinal vessels and perfusion in the macula

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Salvador, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Arnau de Vilanova, Lleida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yau JW, Rogers SL, Kawasaki R, Lamoureux EL, Kowalski JW, Bek T, Chen SJ, Dekker JM, Fletcher A, Grauslund J, Haffner S, Hamman RF, Ikram MK, Kayama T, Klein BE, Klein R, Krishnaiah S, Mayurasakorn K, O'Hare JP, Orchard TJ, Porta M, Rema M, Roy MS, Sharma T, Shaw J, Taylor H, Tielsch JM, Varma R, Wang JJ, Wang N, West S, Xu L, Yasuda M, Zhang X, Mitchell P, Wong TY; Meta-Analysis for Eye Disease (META-EYE) Study Group. Global prevalence and major risk factors of diabetic retinopathy. Diabetes Care. 2012 Mar;35(3):556-64. doi: 10.2337/dc11-1909. Epub 2012 Feb 1. PMID 22301125
- [Background] Garg S, Davis R. Diabetic Retinopathy Screening Update. Clinical Diabetes. 2009;27(4):140-145. doi:10.2337/diaclin.27.4.140
- [Background] van Hecke MV, Dekker JM, Stehouwer CD, Polak BC, Fuller JH, Sjolie AK, Kofinis A, Rottiers R, Porta M, Chaturvedi N; EURODIAB prospective complications study. Diabetic retinopathy is associated with mortality and cardiovascular disease incidence: the EURODIAB prospective complications study. Diabetes Care. 2005 Jun;28(6):1383-9. doi: 10.2337/diacare.28.6.1383. PMID 15920056
- [Background] Rodrigues TM, Marques JP, Soares M, Simao S, Melo P, Martins A, Figueira J, Murta JN, Silva R. Macular OCT-angiography parameters to predict the clinical stage of nonproliferative diabetic retinopathy: an exploratory analysis. Eye (Lond). 2019 Aug;33(8):1240-1247. doi: 10.1038/s41433-019-0401-7. Epub 2019 Mar 22. PMID 30903092
- [Background] Dimitrova G, Chihara E, Takahashi H, Amano H, Okazaki K. Quantitative Retinal Optical Coherence Tomography Angiography in Patients With Diabetes Without Diabetic Retinopathy. Invest Ophthalmol Vis Sci. 2017 Jan 1;58(1):190-196. doi: 10.1167/iovs.16-20531. PMID 28114579